CLINICAL TRIAL: NCT01034332
Title: A Phase II Study With One-cycle Weekly TP-HDFL Followed by Twice Weekly TP-CCRT and Esophagectomy for Locally Advanced Esophageal Cancer
Brief Title: Paclitaxel/Cisplatin/Fluorouracil Followed by Paclitaxel/Cisplatin/Radiotherapy and Esophagectomy for Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chih-Hung Hsu / Department of Oncology, National Taiwan University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200707051M
Record Dates: First submitted 2008-01-07; First posted 2009-12-17 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2009-12

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer; Esophagectomy; Paclitaxel; Induction chemotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- One-cycle induction chemotherapy (Experimental): TP-HDFL, TP-CCRT, Esophagectomy
  Interventions: Procedure: TP-HDFL,TP-CCRT, Esophagectomy

INTERVENTIONS:
Procedure: TP-HDFL,TP-CCRT, Esophagectomy — To determine whether clinical response to one cycle of induction chemotherapy (TP-HDFL) could predict the pathologic complete response to preoperative chemoradiotherapy (TP-CCRT) in patients with locally advanced esophageal cancer.

SUMMARY:
We hypothesize that one-cycle induction chemotherapy may also help to identify chemo-responsive esophageal cancer patients who are highly treatable by definitive CCRT.

DETAILED DESCRIPTION:
We hypothesize that one-cycle induction chemotherapy may also help to identify chemo-responsive esophageal cancer patients who are highly treatable by definitive CCRT.in order to test this hypothesis, we thus propose this phase II clinical study to verify the role of "response to one-cycle induction chemotherapy"in the prediction of pathologic complete response rate to CCRT and tje outcomes for patients with loco-regional esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven esophageal cancer
* Locally advanced diseases T3 N0-1 M0; T1-3 N1 M0; T1-3 or N0-1 M1a
* Age ≥ 18 years old
* ECOG ≤ 2
* Creatinine < 1.5 mg/dl AST, ALT < 2.5 x upper normal limits Bilirubin < 2.0 mg/dl
* WBC > 4,000/μl or ANC>2,000/μl
* Platelet > 100,000//μl
* Informed consent

Exclusion Criteria:

* Invasion to surrounding organs (T4 disease)
* Distant mets (except M1a)
* Prior thoracic irradiation
* Presence of other squamous cell carcinoma of aerodigestive way
* Symptomatic co-morbid diseases
* Previous malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To determine whether clinical response to one cycle of induction chemotherapy (TP-HDFL) could predict the pathologic complete response to preoperative chemoradiotherapy (TP-CCRT | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hung Hsu, M.D, Principal Investigator — National Taiwan University Hospita
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Guo JC, Huang TC, Lin CC, Hsieh MS, Chang CH, Huang PM, Lee JM, Hsu FM, Chia-Hsien Cheng J, Wang HP, Yeh KH, Cheng AL, Hsu CH. Postchemoradiotherapy Pathologic Stage Classified by the American Joint Committee on the Cancer Staging System Predicts Prognosis of Patients with Locally Advanced Esophageal Squamous Cell Carcinoma. J Thorac Oncol. 2015 Oct;10(10):1481-9. doi: 10.1097/JTO.0000000000000651. PMID 26313683